CLINICAL TRIAL: NCT04687397
Title: Investigation of the Behavioral Signs of Consciousness Recovery in Patients With Disorders of Consciousness (DOCSIGNS)
Brief Title: Behavioral Signs of Consciousness Recovery in Patients With Disorders of Consciousness (DOCSIGNS)
Acronym: DOCSIGNS
Status: Completed | Type: Observational
Sponsor: Hospitales Nisa (Other)
Collaborators: Universitat Politècnica de València (Other)
Responsible Party: Principal Investigator, Enrique Noe, Research director, Hospitales Nisa
Other Study IDs: HN19025C73
Record Dates: First submitted 2020-12-17; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Consciousness Disorder; Brain Injuries
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Disorders of consciousness: Patients diagnosed as either in a Vegetative State or in a Minimally Conscious State
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation — Multidisciplinary rehabilitation

SUMMARY:
Precise description of behavioral signs denoting transition from unresponsive wakefulness syndrome/vegetative state (UWS/VS) to minimally conscious state (MCS) or emergence from MCS after severe brain injury is crucial for prognostic purposes. A few studies have attempted this goal but involved either non-standardized instruments, limited temporal accuracy or samples, or focused on (sub)acute patients. The objective of this study is to describe the behavioral signs that led to a change of diagnosis, as well as the factors influencing this transition, in a large sample of patients with chronic disorders of consciousness after severe brain injury.

ELIGIBILITY:
Inclusion Criteria:

* documented medical diagnosis of CRS-R-based diagnosis of UWS or MCS at admission to the neurorehabilitation program

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants were subjects who were diagnosed as with UWS or in a MCS after a brain injury
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline score in the Coma Recovery Scale-Revised until study completion | From inclusion in the study until discharge or death, assessed up to 24 months
  The Coma Recovery Scale-Revised consists of 29 hierarchically organised items divided into 6 subscales addressing auditory, visual, motor, oromotor, communication, and arousal processes.

SECONDARY OUTCOMES:
Change from baseline score in the Functional Independence Measure until study completion | From inclusion in the study until discharge or death, assessed up to 24 months
  The Functional Independence Measure is an 18-item measurement tool that explores an individual's physical, psychological and social function
Change from baseline score in the Disability Rating Scale until study completion | rom inclusion in the study until discharge or death, assessed up to 24 months
  The Disability Rating Scale is an 8-item measure that assesses disability of individuals with moderate to severe traumatic brain injury at a wide range of functional levels from coma through community living

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Noé, Principal Investigator — Hospitales Nisa
Locations (1):
- Servicio de Neurorrehabilitación y Daño Cerebral de los Hospitales NISA, Valencia, Spain